CLINICAL TRIAL: NCT02175108
Title: DIET, ACTIVITY AND MEDICAL CO-MORBIDITIES IN ADOLESCENTS and ADULTS WITH CEREBRAL PALSY: WHAT ARE THE EFFECTS ON THE METABOLIC PROFILE?
Brief Title: Diet and Activity in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Christina Marciniak, Professor, Northwestern University and Attending Physician Shirley Ryan AbilityLab, Northwestern University
Other Study IDs: STU00093759
Record Dates: First submitted 2014-06-22; First posted 2014-06-26 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2016-10

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Adolescents; Adults; Diet; Activity; Metabolic Syndrome
MeSH Terms: conditions — Cerebral Palsy; Motor Activity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to fill a gap in the literature, identify relevant clinical measures, and provide insight into the independent modifiable risk factors of obesity in the CP population with the long-term goal of improving screening, management and prevention of obesity in this at-risk and underserved population.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent and adult subjects 16-89 years with a diagnosis of Cerebral Palsy

Exclusion Criteria:

* Concurrent severe neurologic or other medical diagnosis that is likely to be contributing to the subject's functional impairment, as determined by the study investigators. For example, associated spinal cord injury.
* Subjects with major limb amputations
* Pregnant or lactating females

Ages: 16 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents (16-17) and adults with cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Calories per day | 24 hour dietary recall
  Subjects will complete dietary recall and total calories per day will be calculated
Total saturated fats per day | 24 hour
  24 hour dietary recall will be performed, and total saturated fats ingested over 24 hours will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No